CLINICAL TRIAL: NCT04895254
Title: Colonoscopy Using Motorized Spiral Enteroscope: Prospective Bi-center Study
Brief Title: Colonoscopy Using Motorized Spiral Enteroscope
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Abdulbaqi Al-Toma, Principal investigator, St. Antonius Hospital
Other Study IDs: W2021.204
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Colon Disease
Keywords: Motorized Spiral enteroscopy; colonoscopy
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Motorized spiral Enteroscopy: Consecutive patients with difficult colonoscopies to be enrolled to achieve total colonoscopy using the motorized spiral enteroscope.
  Interventions: Device: Diagnostic colonoscopy; Procedure: Therapeutic colonoscopy

INTERVENTIONS:
Device: Diagnostic colonoscopy — The feasibility of the motorized spiral enteroscope to achieve cecum intubation in difficult colons.
Procedure: Therapeutic colonoscopy — The feasibility of the motorized spiral enteroscope for performing interventions such as polypectomy

SUMMARY:
The new technology of the motorized Spiral enteroscope, originally developed for deep small bowel enteroscopy, might potentially overcome some limitations of standard colonoscopy.

DETAILED DESCRIPTION:
Cecal intubation rate represents a key procedural quality parameter in diagnostic colonoscopy. However, even in experienced hands, a significant percentage of colonoscopies (1.6-16.7%) remain incomplete because of a failure to intubate the cecum. The new technology of the motorized Spiral enteroscope, originally developed for deep small bowel enteroscopy, might potentially overcome some limitations of standard colonoscopy. The study aim was to evaluate the feasibility and safety of motorized Spiral enteroscopy for difficult colonoscopies.

ELIGIBILITY:
Inclusion Criteria:

- Indications for Spiral colonoscopy as a rescue procedure because of incomplete antecedent colonoscopy

Exclusion Criteria:

* Age under 18 years
* Known pregnancy
* Poor health status (ASA classification ≥ 4)
* Contraindication for sedation or standard colonoscopy
* Known coagulopathy (INR ≥ 2.0, platelets < 70 /nl) or anticoagulants other than aspirin
* Medical history of chronic inflammatory bowel disease or suspected bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with failed colonoscopies using the conventional standrad colonoscopy devices.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
evaluate the feasibility of motorized PowerSpiral enteroscopy for difficult colonoscopies | during procedure
  achieving cecum intubation in difficult colons
evaluate the safety of motorized PowerSpiral enteroscopy for difficult colonoscopies | 7 days
  Registering adverse events

SECONDARY OUTCOMES:
Endoscopic mucosal resection | during procedure
  Performing endoscopic mucosal resection on polyps

CONTACTS AND LOCATIONS:
Overall Officials: Abdulbaqi Al-Toma, Ph.D., Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - University Medical Centre Groningen, Groningen
  - St Antonius hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No